CLINICAL TRIAL: NCT00086515
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of the Addition of MK0431 to Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Therapy
Brief Title: Metformin Add-on Study in Patients With Type 2 Diabetes Mellitus (0431-020)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-020; Formally-B0604T2DMT; 2006_411
Record Dates: First submitted 2004-07-02; First posted 2004-07-05 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Glipizide; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sitagliptin 100 mg (Experimental): The Sitagliptin 100 mg group includes patients who were administered once-daily treatment with oral tablets of sitagliptin 100 mg during Phase A (Weeks 0-24) of the treatment period. During Phase B (Weeks 24-104) of the treatment period these patients received once-daily coadministered treatment with oral tablets of sitagliptin 100 mg and glipizide-matched placebo.
  Interventions: Drug: Sitagliptin (MK0431); Drug: Metformin; Drug: Pioglitazone
- Placebo / Glipizide 5 mg (Placebo Comparator): The Placebo/Glipizide 5 mg group includes patients who were administered once-daily treatment with oral tablets of sitagliptin-matched placebo during Phase A (Weeks 0-24) of the treatment period. During Phase B (Weeks 24-104) of the treatment period these patients received once-daily coadministered treatment with oral tablets of sitagliptin-matched placebo 100 mg and glipizide 5 mg which was allowed to be uptitrated, in a blinded fashion, to a maximum dose of 15 mg/day.
  Interventions: Drug: Placebo/Glipizide 5 mg; Drug: Metformin; Drug: Pioglitazone

INTERVENTIONS:
Drug: Sitagliptin (MK0431) — Sitagliptin 100 mg once daily, from Visit 4 through Final Visit, week 104
  Other Names: MK0431; sitagliptin phosphate; Januvia
  Arms: Sitagliptin 100 mg
Drug: Placebo/Glipizide 5 mg — Placebo (to match Sitagliptin 100 mg) from Visit 4 through Visit 8; Glipizide 5 mg from Visit 8, week 24 to Final Visit (Week 104)
  Arms: Placebo / Glipizide 5 mg
Drug: Metformin — Metformin 1500 mg, once daily, from Visit 2 to Final Visit (Week 104)
Drug: Pioglitazone — Pioglitazone 15 mg once daily, for patients not meeting specific glycemic goals during the placebo-controlled treatment period [Phase A], from Visit 5 (Week 6) to Visit 8 (Week 24)
  Other Names: ACTOS

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an investigational drug in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2004-06-30 (Actual); Primary Completion 2005-07-20 (Actual); Study Completion 2007-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Charbonnel B, Karasik A, Liu J, Wu M, Meininger G; Sitagliptin Study 020 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor sitagliptin added to ongoing metformin therapy in patients with type 2 diabetes inadequately controlled with metformin alone. Diabetes Care. 2006 Dec;29(12):2638-43. doi: 10.2337/dc06-0706. PMID 17130197
- [Background] Xu L, Man CD, Charbonnel B, Meninger G, Davies MJ, Williams-Herman D, Cobelli C, Stein PP. Effect of sitagliptin, a dipeptidyl peptidase-4 inhibitor, on beta-cell function in patients with type 2 diabetes: a model-based approach. Diabetes Obes Metab. 2008 Dec;10(12):1212-20. doi: 10.1111/j.1463-1326.2008.00887.x. Epub 2008 May 12. PMID 18476982
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary therapy Period: 13-Jul-2004 through 02-Feb-2007 (for the 2-year Phase A and B periods); 100 study centers worldwide. (46 sites in the United States, 25 sites in 11 countries in Europe, and 29 sites in 13 countries in the rest of the world).
Pre-assignment Details: Patients 18-78 years of age with type 2 diabetes mellitus with inadequate glycemic control (hemoglobin A1C [A1C] ≥7% and ≤10%) on stable doses of metformin (≥1500 mg/day) were eligible to enter the 104-week study.
Period: Phase A (Weeks 0-24)
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg
Started | 464 | 237
Completed | 415 | 192
Not Completed | 49 | 45
Not completed — Adverse Event | 17 | 9
Not completed — Lack of Efficacy | 7 | 13
Not completed — Lost to Follow-up | 4 | 5
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Patient Moved | 2 | 3
Not completed — Protocol-Spec lab discon criteria | 4 | 3
Not completed — Poor compliance | 1 | 0
Not completed — Patient needed prohibited treatment | 0 | 1
Not completed — Personal Circumstance | 1 | 0
Period: Phase A to Phase B Transition Period
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg
Started | 415 | 192
Completed | 391 | 164
Not Completed | 24 | 28
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Patient received Phase A rescue therapy | 16 | 23
Not completed — Protocol-Spec lab discon criteria | 1 | 1
Not completed — Poor compliance | 1 | 0
Not completed — Patient needed prohibited treatment | 1 | 0
Period: Phase B (Weeks 24-104)
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg
Started | 391 | 164
Completed | 201 | 109
Not Completed | 190 | 55
Not completed — Adverse Event | 16 | 10
Not completed — Lack of Efficacy | 94 | 19
Not completed — Lost to Follow-up | 13 | 4
Not completed — Physician Decision | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 15 | 5
Not completed — Patient Moved | 2 | 2
Not completed — Protocol-Specific discontinuation | 5 | 3
Not completed — Protocol-Specific lab discon criteria | 36 | 10
Not completed — Patient Died | 3 | 1
Not completed — Patient needed prohibited treatment | 0 | 1
Not completed — Personal Circumstance | 1 | 0
Not completed — Discontinued in error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg | Total
Number analyzed (Participants) | 464 | 237 | 701
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.4) | 54.7 (9.7) | 54.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 96 | 301
  Male | 259 | 141 | 400
Race/Ethnicity, Customized [Number; unit: participants]
  White | 293 | 159 | 452
  Black | 31 | 14 | 45
  Hispanic | 72 | 28 | 100
  Asian | 49 | 26 | 75
  Other | 19 | 10 | 29
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 170.2 (40.2) | 174.1 (42.0) | 171.5 (41.3)
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] | 8.0 (0.8) | 8.0 (0.8) | 8.0 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 24
Description: A1C is measured as a percent. Thus, this change from
  baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 24, the last non-baseline observed measurement was carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg
Number analyzed (Participants) | 453 | 224
Percent | -0.67 [-0.77 to -0.57] | -0.02 [-0.15 to 0.10]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo / Glipizide 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior AHA status (not on AHA, on monotherapy oral AHA, or on metformin-based oral combination AHA), and baseline A1C; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-0.77 to -0.53]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change from baseline at Week 24 is defined as FPG at
  Week 24 minus FPG at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg
Number analyzed (Participants) | 454 | 226
mg/dL | -16.9 [-21.5 to -12.3] | 8.5 [2.9 to 14.1]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo / Glipizide 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior AHA status (not on AHA, on monotherapy oral AHA, or on metformin-based oral combination AHA), and baseline FPG; Mean Difference (Final Values) = -25.4, 95% CI 2-sided [-31.0 to -19.8]

3. Secondary Outcome: Change From Baseline in 2-hour Post-meal Glucose (PMG) at Week 24
Description: Change from baseline at Week 24 is defined as PMG at Week 24 minus PMG at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg
Number analyzed (Participants) | 387 | 182
mg/dL | -62.0 [-70.2 to -53.8] | -11.4 [-21.7 to -1.0]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo / Glipizide 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior AHA status (not on AHA, on monotherapy oral AHA, or on metformin-based oral combination AHA), and baseline 2-hour PMG; Mean Difference (Final Values) = -50.6, 95% CI 2-sided [-60.5 to -40.8]

ADVERSE EVENTS:
Time Frame: Weeks 0-104
Description: Patients received rescue medication if they met specific glycemic goals. Serious Adverse Events (SAEs) include events that occurred either before or after receiving rescue medication. Other Adverse Events (AEs) only includes those AEs that occurred prior to a patient receiving rescue medication.
Arm/Group | Sitagliptin 100 mg | Placebo / Glipizide 5 mg
Serious Adverse Events (participants affected / at risk) | 54/464 | 21/237
Other Adverse Events (participants affected / at risk) | 210/464 | 124/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=464) | Placebo / Glipizide 5 mg (N=237)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Reflux Oesophagitis (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Death (General disorders) | 2 | 0
Hernia (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 3
Biliary Colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Abdominal Wall Infection (Infections and infestations) | 1 | 0
Bronchitis Acute (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Helicobacter Gastritis (Infections and infestations) | 0 | 1
Infected Epidermal Cyst (Infections and infestations) | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 0
Meningitis Bacterial (Infections and infestations) | 1 | 0
Perirectal Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia Primary Atypical (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Polytraumatism (Injury, poisoning and procedural complications) | 2 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear Cell Carcinoma Of The Kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Follicular Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Pelvic Haematoma (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Finger Amputation (Surgical and medical procedures) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Leriche Syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=464) | Placebo / Glipizide 5 mg (N=237)
Diarrhoea (Gastrointestinal disorders) | 28 | 11
Bronchitis (Infections and infestations) | 26 | 12
Influenza (Infections and infestations) | 37 | 20
Nasopharyngitis (Infections and infestations) | 41 | 16
Upper Respiratory Tract Infection (Infections and infestations) | 49 | 29
Urinary Tract Infection (Infections and infestations) | 22 | 13
Blood Glucose Increased (Investigations) | 8 | 14
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 41
Back Pain (Musculoskeletal and connective tissue disorders) | 33 | 20
Headache (Nervous system disorders) | 20 | 13
Hypertension (Vascular disorders) | 29 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.